CLINICAL TRIAL: NCT04506840
Title: Development of an Educational and Motivational Program to Promote Adherence to Physical Activity and Its Positive Effects in Colorectal Cancer Patients
Brief Title: Physical Activity and Motivation in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Puerta de Hierro University Hospital (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, David González-Cutre Coll, Senior Lecturer, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPS.DGC.01.19
Record Dates: First submitted 2020-07-21; First posted 2020-08-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Physical Exercise; Motivation; Side Effect; Colorectal Cancer
Keywords: Chemotherapy; Exercise; Motivation; Cancer; Well-being
MeSH Terms: conditions — Motor Activity; Colorectal Neoplasms; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Participants will participate in a program of physical exercise during the adjuvant chemotherapy treatment
  Interventions: Other: Physical activity
- Not training group (No Intervention): Participants will not do any intervention, they only will be perform the pre and post-tests.

INTERVENTIONS:
Other: Physical activity — Patients will participate in a program of physical exercise. Resistance training, endurance training, balance and flexibility will be trained with the objective to reduce the side effects of chemotherapy and, in order to improve their quality of life
  Arms: Training group

SUMMARY:
The intervention will be a physical exercise program for colorectal cancer patients during the adjuvant chemotherapy. The exercise program aims on reducing the side effects of the treatment and improving patients' quality of life. In addition, the investigators try to improve endurance and resistance training level, in order to achieve greater physical functionality, survival and general well-being. For this, the investigators will carry out an exercise program based mainly on muscular strength and cardiorespiratory condition. It will last 6 months, with a frequency of 3 days per week, including sessions of 60 minutes. Sessions will consist of three parts: warm-up, main part (endurance and resistance training), and cool down. An individualized and supervised progression of training will take place. The intensity levels will always be adjusted to the initial levels of the participants, always considering their preferences and comfort.

Participants' preferences and exercise history will be considered through an initial interview. Motivational strategies based on self-determination theory will be applied, since it is one of the most used theories in the field of physical exercise. This theory proposes that all people need to feel competent, autonomous and socially related. If these three needs are satisfied, participants will develop more positive (autonomous) forms of motivation, which are related to better consequences such as vitality, enjoyment, quality of life and adherence to physical activity. In addition, motivational strategies will be applied for families and healthcare professionals.

Before starting the program and at the end of it, each eligible patient will be evaluated through:

* Physical activity: strength test of lower and upper limbs, agility test, stress test for cardiorespiratory fitness, physical activity levels, physical condition and body composition.
* Psychological factors: autonomy support, basic psychological need satisfaction, motivation, quality of life, perceived barriers, depression, anxiety, hope, quality of life.
* Clinical parameters: survival rate, side effects, biological factors, treatment delays and planned treatment completion.

DETAILED DESCRIPTION:
Objectives and justification of the project In Spain, cancer is the second cause of death after cardiovascular diseases. However, if it is divided by sex, cancer is the leading cause of death for men and the second cause for women. In recent years there has been an increase in new cases of cancer due to population growth and aging, since 2/3 of cancer patients are older than 65 years. In addition to the impact of this disease on people's quality of life, a high economic cost has been estimated for the health system. For example, the total cost of cancer in 2015 in Spain was 7,168 million euros. This situation represents an important public health problem and therefore implies that research on the factors that can prevent or alleviate this disease should be considered as a priority.

In this regard, there is increasing scientific evidence of the physical and psychosocial benefits of exercise both during and after the treatment of this disease. Nevertheless, only 30-40% of cancer survivors perform the necessary physical activity (PA) recommended by the main medical institutions. In fact, a significant number of patients are obese (33%) and have a low cardiorespiratory condition (45%). Despite this, PA continues to decrease after diagnosis and only 5-10% of patients are physically active during treatment and 20-30% after treatment. Therefore, the development of intervention programs aimed at promoting PA should be a fundamental objective in the fight against cancer and its physical and psychosocial consequences. In this line, our general objective will be to develop a motivation PA program for colorectal cancer patients. Specifically, and considering the gaps existing in the current literature, our general objective is subdivided into the following specific objectives:

* To evaluate the physical, psychosocial and behavioural effects, in the short and medium term, of a physical exercise program in which motivational strategies based on self-determination theory are applied.
* To explore qualitatively the benefits of the physical exercise program, as well as the troubles encountered in its implementation.
* To develop an educational guide and an intervention protocol to encourage motivation and adherence to PA of colorectal cancer patients.

Methodology This study will require a sample size of 34 patients. This calculation was made through the G*power software, by means of an analysis of variance (ANOVA), adjusting the values to p <.05, with a statistical power of 80% and an effect size of 0.5. The patients will be recently diagnosed with colorectal cancer in phases II-III by the oncology service of the Hospital Universitario Puerta de Hierro de Majadahonda. Inclusion criteria include to be between 18 and 75 years old, to be undergoing chemotherapy treatment, and to not have any type of associated pathology that prevents them from performing PA. A intervention with an experimental group and a control group will be conducted, where 17 patients will be assigned to a control group, and 17 patients will perform a supervised motivational exercise program.

Measures Cardiorespiratory fitness. Stress tests adapted to the characteristics of the patients will be performed, both in the type of ergometer and in the protocol. We will use electrocardiographic recording and gas exchange analysis. Aerobic and anaerobic exercise thresholds will be established.

Quality of life. The validated Spanish version of the EORTC-QLQ-CR30 will be used for patients with colorectal cancer.

Body composition. Anthropometries will be carried out to estimate body composition parameters.

Biological parameters. The usual analytics carried out in the hospital during the treatment will be used to check the patient's health status and the side effects of the chemotherapy treatment.

Anxiety. The validated version in Spanish of the Hamilton Anxiety Scale will be used.

Depression. The Spanish version of the Hamilton Depression Scale will be used. Autonomy support. The Spanish version of the Perceived Autonomy Support for Exercise Settings will be used.

Perceived barriers to do PA. This scale will be translated and validated to the Spanish context.

Basic psychological needs in exercise. We will use the Basic Psychological Needs in Exercise Scale.

Basic psychological needs in life. The Spanish version of the Basic Psychological Need Satisfaction and Frustration Scale will be used.

Types of motivation. To measure motivation towards PA, the Behavioural Regulation in Exercise Questionnaire will be for PA levels. The Spanish version of the IPAQ questionnaire will be used. On the other hand, PA will be measured in a direct and objective way through portable GT3X accelerometers.

Design, procedure and data analysis The intervention program will be carried out at the Hospital Universitario Puerta de Hierro of Majadahonda. The program will last 6 months, with three weekly one-hour sessions, and will comply with the recommendations established by the American Cancer Society and the American College of Sports Medicine. The safety precautions and contraindications identified by these institutions for colorectal cancer patients will be especially considered. The program will include aerobic sessions at moderate and vigorous intensities, as well as strength work. Patients will be monitored to model exercise loads individually.

The measurements will be made just before starting the PA program (T1) in the case of the experimental group, at an initial time of the equivalent treatment in the case of the control group. The same measures will be carried out 6 months later (T2). For PA levels, instead of measuring them just after the end of the program, we will wait another month so that patients have been able to recover their usual PA levels after the shock that can mean for them to face the end of our program. In the control group, PA levels will also be evaluated one month after T2. To test the effects of the program, all measurements will be performed 6 months after T2 in both groups (T3).

Additionally, qualitative methodology will be used, so that the 17 patients of the experimental group will be interviewed to know the factors related to their adherence to the PA program and the benefits perceived by them with their participation. Qualitative data collection will be reinforced with field notes compiled in research diaries by observers who will be present during the development of the program. Relatives and health professionals will also be interviewed to learn their perspective regarding the benefits of the program and adherence to it in these patients.

In order to promote adherence to the program and to educate in autonomous PA habits when it ends, motivational strategies based on the self-determination theory will be used. Specific strategies will be developed for this group, based on previous works and educational guides for colorectal cancer patients. The instructor in charge of directing the program will be trained in several sessions to use motivational strategies based on this theory. Once the program is finished, an educational guide of motivational strategies for the promotion of PA in patients with colorectal cancer will be developed and published from the perspective of self-determination theory.

ELIGIBILITY:
Inclusion criteria:

* Being more than 18 years
* Colorectal cancer stage II and III
* Be receiving adjuvant chemotherapy treatment after surgery
* Ecog > 1
* No medical contraindications

Exclusion criteria:

* Have a disability
* Colorectal cancer stage IV
* Presence of metastasis
* Ecog < 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Pre intervention
  Rockport 1-mile walking test
Cardiorespiratory fitness | In the middle of the intervention (at 3 months)
  Rockport 1-mile walking test
Cardiorespiratory fitness | At 6 months after the start of the intervention
  Rockport 1-mile walking test
Cardiorespiratory fitness | One year after the start of the intervention
  Rockport 1-mile walking test
Strength | Pre intervention
  Handgrip strength is a measure of the maximum static force that a hand can squeeze using a dynamometer
Strength | In the middle of the intervention (at 3 months)
  Handgrip strength is a measure of the maximum static force that a hand can squeeze using a dynamometer
Strength | At 6 months after the start of the intervention
  Handgrip strength is a measure of the maximum static force that a hand can squeeze using a dynamometer
Strength | One year after the start of the intervention
  Handgrip strength is a measure of the maximum static force that a hand can squeeze using a dynamometer

SECONDARY OUTCOMES:
Quality of life (physical function, emotional role, social function, cognitive function and symptoms such a fatigue, anorexia, dyspnea, etc) | Pre intervention
  Questionnaire of EORT-QLQ-29 values are assigned between 1 and 4 (1: not at all, 2: a little, 3: quite a bit, 4: a lot) according to the patient's responses to the item, only items 29 and 30 are evaluated with a score of 1 to 7 (1: lousy, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales
Quality of life (physical function, emotional role, social function, cognitive function and symptoms such a fatigue, anorexia, dyspnea, etc) | In the middle of the intervention (at 3 months)
  Questionnaire of EORT-QLQ-29 values are assigned between 1 and 4 (1: not at all, 2: a little, 3: quite a bit, 4: a lot) according to the patient's responses to the item, only items 29 and 30 are evaluated with a score of 1 to 7 (1: lousy, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales
Quality of life (physical function, emotional role, social function, cognitive function and symptoms such a fatigue, anorexia, dyspnea, etc) | At 6 months after the start of the intervention
  Questionnaire of EORT-QLQ-29 values are assigned between 1 and 4 (1: not at all, 2: a little, 3: quite a bit, 4: a lot) according to the patient's responses to the item, only items 29 and 30 are evaluated with a score of 1 to 7 (1: lousy, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales
Quality of life (physical function, emotional role, social function, cognitive function and symptoms such a fatigue, anorexia, dyspnea, etc) | One year after the start of the intervention
  Questionnaire of EORT-QLQ-29 values are assigned between 1 and 4 (1: not at all, 2: a little, 3: quite a bit, 4: a lot) according to the patient's responses to the item, only items 29 and 30 are evaluated with a score of 1 to 7 (1: lousy, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales
Motivation in exercise context | Pre intervention
  Questionnaire BREQ-3 (from 1 to 4 points, being from less autonomous types of motivation to more autonomous types of motivation, based on Self-Determination Theory)
Motivation in exercise context | In the middle of the intervention (at 3 months)
  Questionnaire BREQ-3 (from 1 to 4 points, being from less autonomous types of motivation to more autonomous types of motivation, based on Self-Determination Theory)
Motivation in exercise context | At 6 months after the start of the intervention
  Questionnaire BREQ-3 (from 1 to 4 points, being from less autonomous types of motivation to more autonomous types of motivation, based on Self-Determination Theory)
Motivation in exercise context | One year after the start of the intervention
  Questionnaire BREQ-3 (from 1 to 4 points, being from less autonomous types of motivation to more autonomous types of motivation, based on Self-Determination Theory)
Body composition | Pre intervention
  waist and hip circumference/ waist and hip index
Body composition | In the middle of the intervention (at 3 months)
  waist and hip circumference/ waist and hip index
Body composition | At 6 months after the start of the intervention
  waist and hip circumference/ waist and hip index
Body composition | One year after the start of the intervention
  waist and hip circumference/ waist and hip index
Autonomy support questionnaire | Pre intervention
  Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES). From 1 to 7 points, being more score, more perceived support
Autonomy support questionnaire | In the middle of intervention (at 3 months)
  Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES)Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES). From 1 to 7 points, being more score, more perceived support
Autonomy support questionnaire | At 6 months after the start of the intervention
  Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES)Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES). From 1 to 7 points, being more score, more perceived support
Autonomy support questionnaire | One year after the start of the intervention
  Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES)Support Scale for Perceived Autonomy in Physical Exercise Contexts (PASSES). From 1 to 7 points, being more score, more perceived support
Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) | Pre intervention
  In general life context (from 1 to 5 points)
Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) | In the middle of intervention (at 3 months)
  In general life context (from 1 to 5 points)
Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) | At 6 months after the start of the intervention
  In general life context (from 1 to 5 points)
Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) | One year after the start of the intervention
  In general life context (from 1 to 5 points)
The scale of Basic Psychological Needs in Exercise (BPNES) will be used | Pre intervention
  In exercise context (from 1 to 5 points, being more score, more satisfaction of basic psychological needs)
The scale of Basic Psychological Needs in Exercise (BPNES) will be used | In the middle of intervention (at 3 months)
  (from 1 to 5 points, being more score, more satisfaction of basic psychological needs)
The scale of Basic Psychological Needs in Exercise (BPNES) will be used | At 6 months after the start of the intervention
  (from 1 to 5 points, being more score, more satisfaction of basic psychological needs)
The scale of Basic Psychological Needs in Exercise (BPNES) will be used | One year after the start of the intervention
  (from 1 to 5 points, being more score, more satisfaction of basic psychological needs)
Perceived barriers to physical activity participation questionnaire | Pre intervention
  On this scale, patients are asked how often different barriers (time, pain, cost, fatigue, etc.) have interfered with their participation in physical exercise during cancer treatment.
Perceived barriers to physical activity participation questionnaire | In the middle of intervention (at 3 months)
  On this scale, patients are asked how often different barriers (time, pain, cost, fatigue, etc.) have interfered with their participation in physical exercise during cancer treatment.
Perceived barriers to physical activity participation questionnaire | At 6 months after the start of the intervention
  On this scale, patients are asked how often different barriers (time, pain, cost, fatigue, etc.) have interfered with their participation in physical exercise during cancer treatment.
Perceived barriers to physical activity participation questionnaire | One year after the start of the intervention
  On this scale, patients are asked how often different barriers (time, pain, cost, fatigue, etc.) have interfered with their participation in physical exercise during cancer treatment.
Hope State Questionnaire | Pre intervention
  Scale of hope state to face the disease
Hope State Questionnaire | In the middle of intervention (at 3 months)
  Scale of hope state to face the disease
Hope State Questionnaire | At 6 months after the start of the intervention
  Scale of hope state to face the disease
Hope State Questionnaire | One year after the start of the intervention
  Scale of hope state to face the disease
Physical condition questionnaire | Pre intervention
  International Fitness Scale (IFI)
Physical condition questionnaire | In the middle of intervention (at 3 months)
  International Fitness Scale (IFI)
Physical condition questionnaire | At 6 months after the start of the intervention
  International Fitness Scale (IFI)
Physical condition questionnaire | One year after the start of the intervention
  International Fitness Scale (IFI)
Side effects of the chemotherapy | Pre intervention
  Fatigue questionnaire FACIT
Side effects of the chemotherapy | In the middle of intervention (at 3 months)
  Fatigue questionnaire FACIT
Side effects of the chemotherapy | At 6 months after the start of the intervention
  Fatigue questionnaire FACIT
Side effects of the chemotherapy | One year after the start of the intervention
  Fatigue questionnaire FACIT
Physical activity levels (subjective) | Pre intervention
  International physical activity questionnaire (IPAQ)
Physical activity levels (subjective) | In the middle of intervention (at 3 months)
  International physical activity questionnaire (IPAQ)
Physical activity levels (subjective) | At 6 months after the start of the intervention
  International physical activity questionnaire (IPAQ)
Physical activity levels (subjective) | One year after the start of the intervention
  International physical activity questionnaire (IPAQ)
Physical activity levels (objective) | Pre intervention
  Accelerometer
Physical activity levels (objective) | In the middle of intervention (at 3 months)
  Accelerometer
Physical activity levels (objective) | At 6 months after the start of the intervention
  Accelerometer
Physical activity levels (objective) | One year after the start of the intervention
  Accelerometer
Depression and anxiety | Pre intervention
  The Hospital Anxiety and Depression Scale questionnaire (1-4 scale: never, not very often, sometimes, slmost always, the higher the score worse the result)
Depression and anxiety | In the middle of intervention (at 3 months)
  The Hospital Anxiety and Depression Scale questionnaire (1-4 scale: never, not very often, sometimes, slmost always, the higher the score worse the result)
Depression and anxiety | At 6 months after the start of the intervention
  The Hospital Anxiety and Depression Scale questionnaire (1-4 scale: never, not very often, sometimes, slmost always, the higher the score worse the result)
Depression and anxiety | One year after the start of the intervention
  The Hospital Anxiety and Depression Scale questionnaire (1-4 scale: never, not very often, sometimes, slmost always, the higher the score worse the result)

CONTACTS AND LOCATIONS:
Overall Officials: David González-Cutre Coll, PhD, Principal Investigator — Miguel Hernández University of Elche
Locations (2):
- Spain (2):
  - Universidad Miguel Hernández, Elche, Elche/Alicante
  - Hospital Universitario Puerta de Hierro, Madrid, Majadahonda/Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Alvero Cruz, J. R., Armesilla, M. D. C., Herrero-de-Lucas, A., Riaza, L. M., Pascual, C. M., Manzañido, J. P., … Belando, J. E. S. (2010). Body composition assessment in sports medicine. Statement of Spanish group of kinanthropometry of Spanish federation of sports medicine. Version 2010. Archivos de Medicina del Deporte, 27, 330-344.
- [Background] Arraras JI, Suarez J, Arias de la Vega F, Vera R, Asin G, Arrazubi V, Rico M, Teijeira L, Azparren J. The EORTC Quality of Life questionnaire for patients with colorectal cancer: EORTC QLQ-CR29 validation study for Spanish patients. Clin Transl Oncol. 2011 Jan;13(1):50-6. doi: 10.1007/s12094-011-0616-y. PMID 21239355
- [Background] Courneya, K. S., Friedenreich, C. M., Arthur, K., y Bobick, T. M. (1999b). Understanding exercise motivation in colorectal cancer patients: A prospective study using the theory of planned behavior. Rehabilitation Psychology, 44, 68-84.
- [Background] Courneya, K. S., Friedenreich, C. M., Arthur, K., y Bobick, T. M. (1999a). Physical exercise and quality of life in postsurgical colorectal cancer patients. Psychology, Health, & Medicine, 4, 181-187.
- [Background] Courneya KS, Friedenreich CM, Quinney HA, Fields AL, Jones LW, Fairey AS. Predictors of adherence and contamination in a randomized trial of exercise in colorectal cancer survivors. Psychooncology. 2004 Dec;13(12):857-66. doi: 10.1002/pon.802. PMID 15386794
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Fuller JT, Hartland MC, Maloney LT, Davison K. Therapeutic effects of aerobic and resistance exercises for cancer survivors: a systematic review of meta-analyses of clinical trials. Br J Sports Med. 2018 Oct;52(20):1311. doi: 10.1136/bjsports-2017-098285. Epub 2018 Mar 16. PMID 29549149
- [Background] Garcia DO, Thomson CA. Physical activity and cancer survivorship. Nutr Clin Pract. 2014 Dec;29(6):768-79. doi: 10.1177/0884533614551969. Epub 2014 Oct 21. PMID 25335787
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Lobo A, Chamorro L, Luque A, Dal-Re R, Badia X, Baro E; Grupo de Validacion en Espanol de Escalas Psicometricas (GVEEP). [Validation of the Spanish versions of the Montgomery-Asberg depression and Hamilton anxiety rating scales]. Med Clin (Barc). 2002 Apr 13;118(13):493-9. doi: 10.1016/s0025-7753(02)72429-9. Spanish. PMID 11975886
- [Background] Ng JY, Ntoumanis N, Thogersen-Ntoumani C, Deci EL, Ryan RM, Duda JL, Williams GC. Self-Determination Theory Applied to Health Contexts: A Meta-Analysis. Perspect Psychol Sci. 2012 Jul;7(4):325-40. doi: 10.1177/1745691612447309. PMID 26168470
- [Background] Peddle CJ, Plotnikoff RC, Wild TC, Au HJ, Courneya KS. Medical, demographic, and psychosocial correlates of exercise in colorectal cancer survivors: an application of self-determination theory. Support Care Cancer. 2008 Jan;16(1):9-17. doi: 10.1007/s00520-007-0272-5. Epub 2007 Jun 15. PMID 17569994
- [Background] Rantanen T, Guralnik JM, Foley D, Masaki K, Leveille S, Curb JD, White L. Midlife hand grip strength as a predictor of old age disability. JAMA. 1999 Feb 10;281(6):558-60. doi: 10.1001/jama.281.6.558. PMID 10022113
- [Background] Roman, B., Serra-Majem, L., Hagstromer, M., Ramon, J., Ribas, L., y Sjostrom, M. (2006). International Physical Activity Questionnaire: Reliability and validity in Spain. Medicine and Science in Sports and Exercise, 38, S563. doi:10.1249/00005768-200605001-03214
- [Background] Romero-Elías, M., González-Cutre, D., Beltrán-Carrillo, V. J., y Cervelló, E. (2017). Factors that promote or hinder physical activity participation in patients with colorectal cancer: A systematic review. Psychology, Society, & Education, 9, 201-226.
- [Background] Ruiz-Casado A, Verdugo AS, Solano MJ, Aldazabal IP, Fiuza-Luces C, Alejo LB, del Hierro JR, Palomo I, Aguado-Arroyo O, Garatachea N, Cebolla H, Lucia A. Objectively assessed physical activity levels in Spanish cancer survivors. Oncol Nurs Forum. 2014 Jan 1;41(1):E12-20. doi: 10.1188/14.ONF.E12-E20. PMID 24368248
- [Background] Ryan, R. M., y Deci, E. L. (2017). Self-determination theory: Basic psychological needs in motivation, development, and wellness. New York: Guilford Press.
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Spence RR, Heesch KC, Brown WJ. Colorectal cancer survivors' exercise experiences and preferences: qualitative findings from an exercise rehabilitation programme immediately after chemotherapy. Eur J Cancer Care (Engl). 2011 Mar;20(2):257-66. doi: 10.1111/j.1365-2354.2010.01214.x. PMID 20649808
- [Background] Vlachopoulos, S. P., y Michailidou, S. (2006). Development and initial validation of a measure of autonomy, competence, and relatedness in exercise: The Basic Psychological Needs in Exercise Scale. Measurement in Physical Education and Exercise Science, 10, 179-201.
- [Background] Whistance RN, Conroy T, Chie W, Costantini A, Sezer O, Koller M, Johnson CD, Pilkington SA, Arraras J, Ben-Josef E, Pullyblank AM, Fayers P, Blazeby JM; European Organisation for the Research and Treatment of Cancer Quality of Life Group. Clinical and psychometric validation of the EORTC QLQ-CR29 questionnaire module to assess health-related quality of life in patients with colorectal cancer. Eur J Cancer. 2009 Nov;45(17):3017-26. doi: 10.1016/j.ejca.2009.08.014. Epub 2009 Sep 16. PMID 19765978